CLINICAL TRIAL: NCT05920772
Title: Preventing Smoking Initiation in Adolescents Living in Vulnerable Socioeconomic Situations: a Study Protocol of the KickAsh! Intervention
Brief Title: Process and Effect Evaluation of the KickAsh! Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2023-0366
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Smoking Cigarette; Smoking Tobacco; Smoking; Smoking Prevention
Keywords: Smoking Prevention; RCT-study; Tobacco smoking; Cigarette smoking; Smoking; Smoking initiation; Smoking Start; Smoking onset; adolescents; youth work; low SES; socioeconomic status; vulnerable; evaluation; effect evaluation; process evaluation; co-creation; intervention
MeSH Terms: conditions — Cigarette Smoking; Smoking; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: A two-arm non-randomized controlled trail with a mixed-methods approach will be conducted. Youth social work organisations will be assigned to one of the two groups: 1. one group will receive the intervention (intervention group), 2. another group will not receive the intervention (control group). Measurements will take place in both groups at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A smoking initiation prevention intervention (called KickAsh! intervention) will be implemented in 12 youth social work organisations offering sport and/or recreational activities, during a period of three months (October 2023 to December 2023).Youth workers will act as implementers of the intervention. Approximately 5 youth workers per organisation will participate in the study. Adolescents participating in the youth social work organisations will receive the intervention. Approximately 25 adolescents per organisation will participate in the study.
  Interventions: Behavioral: KickAsh! intervention
- Control group (No Intervention): 12 other youth social work organisations offering sport and/or recreational activities will be allocated to the control group. This group will not receive the KickAsh! intervention. Approximately 5 youth workers per organisation will participate in the study. Approximately 25 adolescents per organisation will participate in the study.

INTERVENTIONS:
Behavioral: KickAsh! intervention — The general aim of the KickAsh! intervention is to prevent smoking initiation in adolescents living in vulnerable socioeconomic situations. The intervention exists of different components concerning smoking prevention. Most components have a direct influence on smoking initiation by affecting several determinants of the adolescents. These components include smoke-free games, mood boards, a smoke-free camp, the Kick some Ash!-challenge and exercises concerning self-efficacy and skills. Yet, some of the components target adolescents by influencing their environment, i.e. smoking policy in the organisation and youth workers as role models. All components are developed using a combination of theoretical methods to change or influence these determinants or environmental factors.
  Arms: Intervention group

SUMMARY:
The goal of this evaluation study is to evaluate the KickAsh! intervention, an intervention aiming to prevent smoking initiation in adolescents living in vulnerable socioeconomic situations. This intervention will be implemented in youth social work organisation that offer sport and/or recreational activities for these adolescents. Youth workers will act as implementers of the intervention.

The main aim of this study is to evaluate the effect of the intervention, whether it does or does not produce change in the smoking initiation behaviour of adolescents (= effect evaluation). Secondly, the study aims to evaluate the implementation process to generate more understanding concerning why the intervention does or does not produces change. Therefore, it will be investigated how the intervention was implemented, what exactly was implemented, in which context the intervention was implemented... (= process evaluation)

For the effect evaluation adolescents will be asked to fill in a questionaire at three time points. For the process evaluations interviews and focus groups will be organised with the adolescents and youth workers respectively.

Two groups will participate to this study: one group existing of organisations where the intervention will be implemented (=intervention group), and one group where the intervention will not be implemented (= control group).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 15 years old
* Participate in activities offered by a youth social work organisation during the implementation period
* Have sufficient understanding of the Dutch language

Exclusion Criteria:

* Not participating in a youth social work organisation

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in smoking initiation behaviour at 3 months | From enrollment to the end of intervention implementation at 3 months
  Smoking initiation will be measured following MUSICA: the Model of Unplanned Smoking Initiation of Children and Adolescents. In addition, two questions will be asked concerning smoking frequency in the past month and in adolescents life. Smoking onset age and smoking intention in the following year an d the future are also questioned.
Change in smoking initiation behaviour at 6 months follow-up | From end of intervention implementation to follow-up measurement after 6 months
  Smoking initiation will be measured following MUSICA: the Model of Unplanned Smoking Initiation of Children and Adolescents. In addition, two questions will be asked concerning smoking frequency in the past month and in adolescents life. Smoking onset age and smoking intention in the following year an d the future are also questioned.

SECONDARY OUTCOMES:
Change in attitude towards smoking at 3 months | From enrollment to the end of intervention implementation at 3 months
  8 items will be assessed: 4 items for cognitive and 4 items for emotional (dis)advantages of smoking. Adolescents will have to answer using a five-point likert scale.
Change in attitude towards smoking at 6 months follow-up | From end of intervention implementation to follow-up measurement after 6 months
  8 items will be assessed: 4 items for cognitive and 4 items for emotional (dis)advantages of smoking. Adolescents will have to answer using a five-point likert scale.
Change in self-efficacy concerning smoking at 3 months | From enrollment to the end of intervention implementation at 3 months
  Self-efficacy will be measured via 6 questions measuring the ability to resist smoking in several situations (5-point likert scale). These questions will be linked to 6 coping plan items.
Change in self-efficacy concerning smoking at 6 months follow-up | From end of intervention implementation to follow-up measurement after 6 months
  Self-efficacy will be measured via 6 questions measuring the ability to resist smoking in several situations (5-point likert scale). These questions will be linked to 6 coping plan items.
Change in social influence concerning smoking at 3 months | From enrollment to the end of intervention implementation at 3 months
  Social influence will be measured by assessing perceived social norm (7 questions determining the perceptions of important people in the adolescent's environment) and social pressure (7 items determining the pressure felt by adolescents by the same important people). Both via a 5-point likert scale.
Change in social influence concerning smoking at 6 months follow-up | From end of intervention implementation to follow-up measurement after 6 months
  Social influence will be measured by assessing perceived social norm (7 questions determining the perceptions of important people in the adolescent's environment) and social pressure (7 items determining the pressure felt by adolescents by the same important people). Both via a 5-point likert scale.
Impact of context on study effects during implementation | From enrollment to the end of intervention implementation at 3 months
  Context of the youth social work organisations will be analysed through interviews and focus groups with respectively adolescents and youth workers.
Mechanisms of impact concerning the delivered intervention | From enrollment to the end of intervention implementation at 3 months
  Mechanisms of impact will be analysed through interviews and focus groups with respectively adolescents and youth workers.
Impact of implementation process on the delivered intervention | From enrollment to the end of intervention implementation at 3 months
  Implementation process (how was it delivered, feasibility, barriers and facilitators...) will be analysed through interviews and focus groups with respectively adolescents and youth workers.
Impact of delivered intervention on the study effects | From enrollment to the end of intervention implementation at 3 months
  What is delivered (fidelity, reach, dose, adaptations) will be analysed through interviews and focus groups with respectively adolescents and youth workers.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté Verloigne, Prof. dr., Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - University Ghent, Ghent, Oost-Vlaanderen
  - University Ghent, Ghent

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised data might be shared with researchers from the research group Health Promotion (Ghent University) for secondary data analyses or teaching purposes. However, participants must re-consent for the use of their data in a new research project and domain.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data collection will take place from September 2023 until July 2024, afterwards data will be pseudonymised and shared. Pseudonymised data will be available for the research group Health Promotion (Ghent University) for at least 10 years, to support an open science view.
Access Criteria: Everyone who possess the URL and login details can access the pseudonymised data files (which are stored on a protected data base from Ghent University).

REFERENCES:
- [Background] Leta K, Lauwerier E, Willems S, Vermeersch S, Demeester B, Verloigne M. Smoking prevention within social work organizations: a qualitative study about youngsters' and youth workers' perceptions. Health Promot Int. 2023 Jun 1;38(3):daad047. doi: 10.1093/heapro/daad047. PMID 37202340
- [Derived] Demeester B, Verloigne M, Willems S, Leta K, Lauwerier E. Preventing smoking initiation in adolescents living in vulnerable socioeconomic conditions: Study protocol of the KickAsh!-intervention. Scand J Public Health. 2025 May;53(3):330-341. doi: 10.1177/14034948241236232. Epub 2024 Mar 13. PMID 38481024